CLINICAL TRIAL: NCT03495700
Title: Lateral Sinus Floor Elevation in Implant Therapy: A Randomized Controlled Clinical Trail: L-PRF Block Compared With DBBM.
Brief Title: Lateral Sinus Floor Elevation in Implant Therapy.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Dentsply International (Industry)
Responsible Party: Principal Investigator, Drs. Simone Cortellini, Clinical and Research Associate, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Cortellini60095
Record Dates: First submitted 2018-03-19; First posted 2018-04-12 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Edentulous; Alveolar Process, Atrophy
MeSH Terms: conditions — Mouth, Edentulous; Atrophy

STUDY DESIGN:
Intervention Model Description: This study is designed as a randomized controlled clinical trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- L-PRF block (Experimental): For the test group the sub-sinus cavity will be filled with L-PRF block and the window will be closed with L-PRF membranes.
  Eight tubes (9 ml) of venous blood will be collected from the patients. For 6 tubes (red cap) a 12 min centrifugation at 2700 rpm/408g RCF will be followed. Two tubes (white cap) will be centrifuged (IntraSpin, Intra-Lock, Florida, USA) for 3 minutes only to form the Liquid Fibrinogen.
  The L-PRF clots will be removed from the tubes using surgical tweezers. The clots will be thereafter gently compressed into membranes using a sterile metal box (Xpression, Intra-Lock, Florida, USA).
  To prepare the L-PRF Block, L-PRF membranes will be cut into small pieces and mixed with DBBM (Bio-Oss Small particles, Geistlich AG, Wolhusen, Switzerland). The Liquid Fibrinogen will be added to the homogeneous mix, and stirred gently for ± 10 seconds while shaping it to the L-PRF block
  Interventions: Procedure: L-PRF block
- DBBM (Active Comparator): For the control group the sub-sinus cavity will be filled with deproteinized bovine bone mineral (DBBM). The product used will be a xenograft (Bio-Oss Small particles, Geistlich AG, Wolhusen, Switzerland). The window will be closed with a collagen membrane (Bio-Gide, Geistlich AG, Wolhusen, Switzerland).
  Interventions: Procedure: DBBM

INTERVENTIONS:
Procedure: L-PRF block — The use of the L-PRF block as graft material for sinus augmentation procedure will be analysed
  Arms: L-PRF block
Procedure: DBBM — The use of bovine xenograft will be analysed
  Arms: DBBM

SUMMARY:
The L-PRF block is a combination of bone substitute with L-PRF. The use of a L-PRF block in bone augmentation therapies could enhance and improve bone regeneration.

The primary objective of this study is to evaluate if the use of autologous leukocytes and platelet rich fibrin accelerate and promotes bone regeneration in the sinus in comparison with the standard sinus lift procedure procedure.

DETAILED DESCRIPTION:
This is a randomized controlled clinical trial. A total of 24 patients, needing sinus lift with lateral window technique (L), will be enrolled. All patients have to fulfil all of the inclusion and none of the exclusion criteria. The trial will comprise 8 visits. Written informed consent will be obtained prior to any examination carried out for study purposes. Randomization will be performed using sealed, sequentially numbered, opaque envelopes containing treatment allocation.

Under local anaesthesia, the required L will be performed. Once the blood extraction is done the surgery can start following the normal procedure for the lateral approach of sinus floor elevation. Once the preparation of the sinus floor elevation is done the randomization envelopes will be open and the selected treatment will be applied. For the test group the sub-sinus cavity will be filled with L-PRF block and the window will be closed with L-PRF membranes. For the control group the sub-sinus cavity will be filled with only DBBM and the window will be closed with a collagen membrane. Afterwards suturing will be conducted and a CBCT will be taken for control and observation.

After 6 months the subjects return for a check-up of the healing process. A CBCT will be taken to assess the bone regeneration. Implant surgery will be discussed.

With a crestal incision the implant site will be exposed. A trephine bur of 3 mm in diameter will be use to obtain a biopsy of the test or control site. This will result in a biopsy sample of the healed site. At the exact same location of the biopsy the drilling will be performed according to implant protocol and the implant will be placed and ISQ values will be recorded. Follow-up will be till 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent
* Need for L and oral implant placement.
* RBH <4mm
* RBH >4mm, but no T possible (due to anatomy)

Exclusion Criteria:

* Unlikely to be able to comply with the study procedures, as judged by the investigator
* Untreated periodontal disease
* Unfavorable plaque control
* Known or suspected current malignancy
* History of chemotherapy within 5y prior to study
* History of radiation on the head and neck region
* History of other metabolic bone diseases
* Need for systemic corticosteroids
* Current or previous use of intravenous/oral bisphosphonates
* Present alcohol and/or drug abuse
* Involvement in the planning and conduct of the study
* Psychiatric disorders which do not allow a normal treatment outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-03-19 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Volumetric bone regeneration | 6 months
  Amount of bone formation after lateral sinus floor elevation scored at implant placement and after loading, measured on CBCT images. Following a healing period of 5 and 18 months a CBCT will be taken to evaluate the height and width of the newly formed bone and compare it to the initial CBCT. A 3-D volumetric analysis of the amount of gained bone is conducted with MeVisLab software.
Linear bone regeneration | 6 months
  Amount of bone formation after lateral sinus floor elevation scored at implant placement and after loading, measured on CBCT images. Following a healing period of 5 and 18 months a CBCT will be taken to evaluate the height and width of the newly formed bone and compare it to the initial CBCT. 2-D measurements will be performed.

SECONDARY OUTCOMES:
Implant stability based on resonance frequency | 4 months
  Measurements of the implant stability via Osstell ISQ implant stability device. At implant placement and abutment connection a measurement via Osstell ISQ implant stability device will be done.
Histology: evaluation of bone biopsy at implant site | 6 months
  Histological evaluation of a biopsy at implant site. Biopsy samples will be analysed histological to evaluate differences between both groups (density of bone, trabecular thickness, new bone)

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided